CLINICAL TRIAL: NCT06743399
Title: The Effect of Evidence-Based Care Bundle Applıcatıon in the Prevention of Peripheral Venous Catheter-Related Phlebitis Development
Brief Title: Care Bundle Applıcation in the Prevention of Phlebitis
Acronym: Non-randomized
Status: Completed | Type: Observational
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Tuğba DOST, Assist. Prof, Karamanoğlu Mehmetbey University
Other Study IDs: Karamanoglu Mehmetbey U
Record Dates: First submitted 2024-12-03; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: All Patients with Peripheral Venous Catheters
Keywords: Peripheral venous catheterization.; phlebitis; nursing,; care bundle,; experimental study.
MeSH Terms: conditions — Phlebitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Experimental Group: The experimental group included patients who received training, follow-up care, and the care bundle. Patients provided consent, completed demographic forms, and their PVC applications were assessed daily using the "Phlebitis Care Bundle Follow-up Form." Full compliance with all care bundle parameters was required, and non-compliant patients were excluded. Nurses received feedback, and phlebitis symptoms were recorded daily. Monitoring continued until catheter removal or patient discharge. Data collection took place daily from 09:00-12:00, lasting about 2.5 hours.

SUMMARY:
This study was designed as a non-randomized controlled trial, comprising both experimental and control groups, to evaluate the efficacy of an evidence-based care bundle in preventing the development of peripheral venous catheter-related phlebitis. The study was conducted at a goverment hospital, specifically within the Internal Diseases/Injury Care and Neurology/Neurosurgery Departments. Data collection involved the use of several instruments: the Nurse Descriptive Characteristics Form, the Patient Demographic and Clinical Information Form, the Phlebitis Evaluation Scale, and the Bundle Care Clinical Follow-up Form. Patients in the control group received standard care as per the clinic's protocols, while nurses were trained in the principles of care, phlebitis management, and the implementation of care bundles. Patients in the experimental group received care according to the evidence-based care bundle prepared for this study. Statistical analysis of the data was performed using Chi-square and Fisher's Exact tests. Care bundle application was found to be effective in decreasing the rate of PVC-related phlebitis development.

DETAILED DESCRIPTION:
Peripheral venous catheterization (PVC) is a procedure that involves the insertion of a cannula into the lumen of a vein through the patient's skin. It is among the most commonly performed invasive nursing interventions in hospitalized patients. PVC is utilized at various stages of care for approximately 80% of patients during their hospital stay, serving multiple purposes, including meeting their fluid requirements, maintaining fluid-electrolyte balance, administering pharmacological treatments, transfusing blood and blood products, providing total parenteral nutrition (TPN), ensuring vascular access, and monitoring hemodynamic parameters.

When performed appropriately, PVC is a valuable procedure that can be lifesaving for patients. However, improper application or inadequate catheter care can lead to significant local complications, such as infiltration, extravasation, and hemorrhage, as well as systemic complications, including embolism, infection, and circulatory overload. Among these complications, phlebitis, characterized by pain and tenderness along the vein due to inflammation of the intima layer, is particularly common. A variety of factors contribute to the development of phlebitis. Individual factors include advanced age, gender, neutropenia, malnutrition, cancer, cardiovascular diseases, immunosuppression, existing infections, diabetes, smoking, confusion, dementia, and impaired consciousness. Mechanical factors involve the type and size of catheter, the duration of catheter placement, and the anatomical site of insertion. Chemical factors encompass the pH and osmolarity of fluids, as well as the introduction of antiseptic solutions into the vein. Additionally, procedural factors such as the frequency of set changes, maintenance of aseptic conditions, care of the catheter site, and the type of dressing materials used also play a significant role in the incidence of phlebitis.

The Infusion Nurses Society (INS) and the Infusion Nurses Association (INA) recommend that the incidence of phlebitis in a specified patient population should remain below 5%. However, the literature indicates that the incidence of phlebitis varies widely, with reported rates ranging from 1.25% to 80%. In specific studies conducted in our country, the incidence of phlebitis has been reported to be considerably higher, ranging from 17% to 67%. This variability may be attributed to differences in healthcare practices, infection control measures, and patient demographics.

Phlebitis is a common but preventable complication in clinical practice. Enhancing the quality of care to prevent such complications has led to the prominence of care bundles, which are structured sets of clinical practices aimed at preventing specific complications or improving particular clinical outcomes. The care bundle approach entails the simultaneous and complete implementation of scientifically validated practices, applied in a step-by-step manner. Resarch indicates that the application of these practices as a cohesive whole yields better outcomes compared to their individual application. Each component of a care bundle should consist of commonly accepted practices that are supported by evidence, preferably derived from randomized controlled trials classified at evidence levels I and II. Maintaining high compliance with care bundle protocols enhances their effectiveness and overall quality of care, ultimately contributing to reductions in both mortality and morbidity.

Researches that the application of care bundles leads to improved clinical outcomes. Studies have been demonstrated implementation of care bundles significantly reduces the incidence of ventilator-related pneumonia (VRP) and central venous catheterization-related blood circulation infections (CVCR-BCI).

Null Hypothesis (H0) = The application of evidence-based care bundles does not affect the prevention of the development of peripheral venous catheter-related phlebitis.

Alternative Hypothesis (H₁) = The application of evidence-based care bundles positively affects the prevention of peripheral venous catheter-related phlebitis.

In this study, a non-randomized controlled trial was designed and executed, incorporating both control and experimental groups. The methodology followed the guidelines of the Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) guidelines for case-control studies.

ELIGIBILITY:
Inclusion Criteria:

* Received inpatient treatment for at least 72 hours Internal Medicine/Wound Care Clinic and Neurology/Neurosurgery clinics,
* PVK is applied in specified clinics,
* No existing phlebitis,
* No bleeding, clotting or circulatory disorders (learned from patient records),
* Not receiving immunosuppressive, chemotherapy and radiotherapy treatments,
* 18 years and above,
* Patients who volunteered to participate in the study were included in the study.

Exclusion Criteria:

* Transferred to another clinic,
* Died during the research process,
* (For experimental group patients) Failure to fully comply with the care package,
* Patients who wanted to leave the study after agreeing to participate in the study were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in the study are individuals who have received inpatient treatment for at least 72 hours in the Internal Medicine/Wound Care Clinic and Neurology/Neurosurgery clinics of Karaman Training and Research Hospital, Turkiye have undergone PVK application in the specified clinics, do not have existing phlebitis, have no bleeding, clotting, or circulatory disorders (as determined from patient records), are not receiving immunosuppressive therapy, chemotherapy, or radiotherapy, are aged 18 or older, and have voluntarily agreed to participate in the study.
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Phlebitis Care Bundle Clinical Follow-up Form | The evaluation took an average of 6 months until the completion of the study.
  This form was developed to track and record the daily application of nursing interventions from the evidence-based care bundle designed to prevent the development of PVC-related phlebitis.
Phlebitis Evaluation Scale | The evaluation took an average of 6 months until the completion of the study.
  The Phlebitis Evaluation Scale developed by the Intravenous Nursing Society (2006) was used to assess phlebitis symptoms in the area where PVC was placed. The scale ranges from 0 to 4, where 0 indicates no symptoms, 1 indicates redness and/or pain in the catheter entry point, 3 indicates redness, pain, and/or edema at the catheter entry point, red line, and palpation of the vein as a cable, and 4 includes symptoms such as redness, pain, and/or edema at the catheter entry point, red line, palpation of the vein as a cable, being longer than 2.5 cm, and purulent drainage. The researcher observes the PVC area and determines the degree of phlebitis.
Peripheral Venous Catheter Observation | The evaluation took an average of 6 months until the completion of the study.
  The form, created by the researcher, was designed to daily record the phlebitis symptoms and degree included in the Phlebitis Evaluation Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Karamanoğlu Mehmetbey Üniversitesi Sağlık Hizmetleri MYO, Karaman, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code